CLINICAL TRIAL: NCT04947384
Title: Pulmonary Vascular Hemodynamics Before and After Mitral Valve Procedures
Status: Withdrawn | Type: Observational
Why Stopped: PI moved to a different institution. Low enrollment rate.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Ahmed Zaky, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: IRB-300006686; UAB (Other: Anesthesiology)
Record Dates: First submitted 2021-05-18; First posted 2021-07-01 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with moderate mitral valve disease, undergoing interventions: Patients with established WHO-2 diagnosis of PH undergoing open and interventional mitral valve procedures.
  Interventions: Diagnostic Test: To discern micro-RNA specific for right and left heart induced PH
- Patients undergoing mitral valve interventions without pulmonary hypertension: Patients with no PH undergoing open and interventional mitral valve procedures. This group will serve as a control.
  Interventions: Diagnostic Test: To discern micro-RNA specific for right and left heart induced PH
- Patients with precapillary pulmonary hypertension scheduled for right heart catheterization: Patients with established diagnosis of WHO-1-4 groups of PH undergoing right heart catheterization. This group will serve as a control.
  Interventions: Diagnostic Test: To discern micro-RNA specific for right and left heart induced PH

INTERVENTIONS:
Diagnostic Test: To discern micro-RNA specific for right and left heart induced PH — While undergoing other procedures, the investigators will be collecting a total of three blood samples. The first sample will be obtained on arterial cannulation before the initiation of the intervention, the second sample will be collected upon the end of the procedure prior to leaving the procedure room, and the third sample will be collected on the day of discharge from the hospital.

SUMMARY:
The objective of this proposal is to study circulating and echocardiographic markers of pulmonary vascular and right ventricular remodeling in patients with a WHO-2 diagnosis of pulmonary hypertension after mitral valve procedures. The investigators are proposing the study will be impactful for the early detection and prediction and of residual pulmonary hypertension (PH) that would otherwise be undetected and fatal with no curative treatment.

DETAILED DESCRIPTION:
The investigators will enroll 3 groups: Group 1: Patients with established WHO-2 diagnosis of PH undergoing open and interventional mitral valve procedures. Group 2: Patients with no PH undergoing open and interventional mitral valve procedures. Group 3: Patients with established diagnosis of WHO-1-4 groups of PH undergoing right heart catheterization. Groups 2 and 3 will serve as controls. All procedures will be performed at the main UAB Hospital cardiac surgical operating rooms and at the cardiac angiographic suites. The investigators will collect a total of 3 blood samples; the first sample will be obtained on arterial cannulation before the initiation of the intervention, the second sample will be collected upon the end of the procedure prior to leaving the procedure room, and the third sample will be collected on the day of discharge from the hospital. A comprehensive echocardiogram at the 3 corresponding time points of the blood samples obtained; before, and after the intervention and before discharge.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years/old

Exclusion Criteria:

* Patients with ejection fraction (EF) < 35%
* Patients with severe tricuspid valve regurgitation
* Transplant patients
* Patients scheduled for ventricular assist devices
* Patients with a diagnosis of heart failure with preserved ejection fraction
* Any aortic valvular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing mitral valve procedures at the University of Alabama at Birmingham main hospital
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Biomarker analysis | From baseline through one year
  observation of tissue anomalies in target patients

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Zaky, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham, Birmingham, Alabama, United States